CLINICAL TRIAL: NCT04935944
Title: Effect of Variations of Field of View (FOV) and Milliampere (mA) on Metal Artifacts Produced by Dental Implants in Cone Beam Computed Tomography Image Quality. (In-vitro Study)
Brief Title: Effect of FOV and mA on Metal Artifacts on CBCT
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Roshan Adel Ahmed Elsayed, Master student in Cairo university, Cairo University
Other Study IDs: ORAD-CU-2021
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Metal Artifacts; Implant

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tube potential difference (FOV): Using different FOV and mA values of the CBCT machine
  Interventions: Radiation: CBCT radiation

INTERVENTIONS:
Radiation: CBCT radiation — CBCT scanning

SUMMARY:
The aim of this study is to evaluate the effect of exposure parameters as milliampere (mA) and field of view (FOV) in CBCT on metal artifact of dental implant.

DETAILED DESCRIPTION:
Cone Beam Computed Tomography (CBCT) is considered an important valuable imaging technique in the diagnosis and treatment planning in oral and maxillofacial surgery as well as implant dentistry by means of three dimensional images which provide extra information about the buccolingual dimension of the alveolar bone with more details for bone anatomy and inclination.

To make an accurate diagnosis and treatment planning, we have to obtain images with more details and good resolution and quality which could be achieved by CBCT. However, there are some issues in scanned areas that can affect their quality such as presence of metals (metallic restorations, orthodontic appliances, dental implants, crowns) which result in artifacts which can be considered as an important cause of poor image quality which will lead to poor diagnosis.

There are many types of artifacts which can be observed on CBCT images. Beam hardening artifact is considered a common one which occurs when an x-ray beam comprised of polychromatic energies passes through an object, resulting in selective attenuation of lower energy photons. The effect is conceptually similar to a high-pass filter, in that only higher energy photons are left to contribute to the beam and thus the mean beam energy is increased ("hardened").

ELIGIBILITY:
Inclusion Criteria:

* Bio models of jaw with dummy implant.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Using different dry human mandibles with dummy implants.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-03-09 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Dental implant linear measurement | 2 months
  The implant length and width in millimeters will be assessed in the presence of the artifacts with change in the potential difference of FOV and mA

CONTACTS AND LOCATIONS:
Overall Officials: Noha Issa, Associate Prof, Study Director — Cairo University
Locations (1):
- Roshan Adel, Cairo, Giza Governorate, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-15): https://cdn.clinicaltrials.gov/large-docs/44/NCT04935944/Prot_SAP_001.pdf